CLINICAL TRIAL: NCT05505123
Title: Comparison of Sevoflurane and Propofol for Botulinum Toxin Injection in Cerebral Palsy Children: A Prospective, Randomized Trial
Brief Title: Sevoflurane and Propofol for Botulinum Toxin Injection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YUMC 2022-07-038-001
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; sevoflurane; propofol; deep sedation; botulinum toxin
MeSH Terms: conditions — Cerebral Palsy | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane (Experimental): induction and maintenance with sevoflurane
  Interventions: Drug: Sevoflurane
- propofol (Experimental): induction and maintenance with propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — induction and maintenance with sevoflurane for deep sedation
  Other Names: sevoflurane group
  Arms: sevoflurane
Drug: Propofol — induction and maintenance with propofol for deep sedation
  Other Names: propofol group
  Arms: propofol

SUMMARY:
The investigators would like to compare clinical features (onset, duration, emergence time), efficacy of deep sedation (successful completion of procedure), safety (adverse events) and caregiver's satisfaction for sedation when used propofol and sevoluflurane for deep sedation in 3-11 year old pediatric patients with spastic cerebral palsy receiving botulinum toxin injection.

DETAILED DESCRIPTION:
Cerebral palsy is the most common cause of spastic movement disorders in children. Because botulinum toxin blocks nerve transmission and relieves excessive muscle contraction, it is widely used in the treatment of spastic movement disorders in children with cerebral palsy. Botulinum toxin should be injected into the motor end plate of the neuromuscular junction to increase the therapeutic effect and reduce the immune resistance, and side effects. However, it is difficult for pediatric patients to maintain an immobile posture due to fear of the procedure and injection pain. Moreover, even if a patient with cerebral palsy has the will to maintain an immobile posture through preoperative interviews and prior education, it is not easy to control body movements by themselves due to stiffness.

Botulinum toxin injection is a simple procedure, so the procedure time is very short, usually 5-10 minutes. Therefore, it was performed while maintaining spontaneous breathing without an invasive airway maintenance device (e.g., using a neuromuscular blocker and inserting an endotracheal tube or superior laryngeal airway maintainer), unless difficult airway management is anticipated. It is important to provide a deep sedation during the procedure and then to allow for a rapid recovery of consciousness when the drug is stopped after the procedure. Therefore, in clinical practice, intravenous anesthetic such as propofol or inhaled anesthetic such as sevoflurane, both are short-acting drugs, are administered to induce and maintain deep sedation.

When using propofol, the drug can be administered through the intravenous route secured in advance in all patients before sedation or anesthesia, so sedation can be quickly induced without patient cooperation. It has the advantage of being able to restore consciousness without emergence delirium during awakening. However, when propofol is administered intravenously, pain may occur, respiration and cardiovascular depression may be compromised. In addition, because pharmacokinetic model equipment that can monitor the effect site (brain) drug concentration in real time is not universally used in children, the propofol dosage is often adjusted according to the patient's response which leads to a risk of being administered excessively or inadequately.

When using sevoflurane, it can induce sedation without injection pain. When the drug administration is stopped after the procedure, the drug can be eliminated through the patient's exhalation, which leads to rapid recovery of consciousness. Through anesthetic circuit, the concentration of the drug administered to and removed from the patient can be measured in real time, so it is easy to adjust the drug administration dose. Sevoflurane has the advantage of having some muscle relaxation effect in contrast to propofol. However, since sedation is induced only when the drug is inhaled through spontaneous respiration, patient cooperation is required. The frequency of occurrence of delirium and nausea/vomiting during emergence of sevoflurane is higher than that of propofol.

However, to date, no studies directly comparing the clinical aspects (safety, effectiveness, recovery, adverse events) and satisfaction with sedation of propofol and sevoflurane, for deep sedation during botulinum toxin injection in children with cerebral palsy, have not been reported. Therefore, the investigators would like to compare clinical features (onset, duration, emergence time), efficacy of deep sedation (successful completion of procedure), safety (adverse events) and caregiver's satisfaction for sedation when used propofol and sevoluflurane for deep sedation in 3-11 year old pediatric patients with spastic cerebral palsy receiving botulinum toxin injection.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy (ages 3-11)

Exclusion Criteria:

① Obestity : Body Mass Index of 30 kg/m2 or more

* Heart disease : NYHA class >2

  * Laryngomalacia

    * Acute upper respiratory disease or asthma ⑤ Gastroesophageal reflux disease ⑥ Allergy to general anesthetics and drugs planned for use in this study

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
emergence time | up to 1 hour
  1 hour from discontinuation of drug administration to regain of consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee Jung, M.D.,PhD, Principal Investigator — Yeungnam University Hospital
Locations (1):
- Yeungnam University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No